CLINICAL TRIAL: NCT05349084
Title: PET MYOCARDIAL Blood Flow Comparison to Coronary CTA and CT-FFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201904112
Record Dates: First submitted 2022-04-11; First posted 2022-04-27 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET-cCTA-cFFR (Other): patients presenting with stable angina and a moderate pretest likelihood for CAD who are already scheduled to undergo ICA for the clinical indication of angina will be recruited to undergo PET-cCTA-cFFR
  Interventions: Diagnostic Test: PET-cCTA-cFFR

INTERVENTIONS:
Diagnostic Test: PET-cCTA-cFFR — patients presenting with stable angina and a moderate pretest likelihood for CAD who are already scheduled to undergo ICA for the clinical indication of angina will be recruited to undergo PET-cCTA-cFFR

SUMMARY:
The broad, long-term objective of this pilot study is to develop an optimal, clinically usable, non-invasive evaluation of Coronary Artery Disease (CAD) in the setting of stable angina which provides both anatomic and functional information.

Patients already scheduled to undergo Invasive coronary catheterization (ICA) for the clinical indication of angina will be recruited to under go stress-rest Positron Emission Tomography-Coronary CT Angiography-Fractional Flow Reserve (PET-cCTA-cFFR)

DETAILED DESCRIPTION:
This is a single cohort, technology assessment study. Thirty-five patients presenting with stable angina and a moderate pretest likelihood for CAD who are already scheduled to undergo invasive coronary angiography (ICA) for the clinical indication of angina will be recruited to undergo a cCTA examination with FFR followed immediately by regadenoson stress-rest PET on the same PET/CT scanner.

Sensitivity, specificity, NPV, PPV of CTA-cFFR will be obtained using the reference standard of standard of care ICA with FFR for each epicardial coronary artery.

Segmental stress PET MBF will be compared to presence or absence of a coronary artery stenosis ≥ 50% diameter on CCTA and ICA.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age, of either sex
* Patients presenting with stable angina and a moderate pretest likelihood for CAD and scheduled to undergo ICA for the clinical indication of angina. Subjects will undergo this study within 45 days prior to the cardiac catheterization. This study can also be performed 45 days after the cardiac catheterization if the patient had no interventions.

Exclusion Criteria:

* Prior history of stenting, coronary artery bypass graft surgery, or myocardial infarction, unstable angina, atrial fibrillation, second or third degree atrioventricular block, class IV heart failure
* Iodine allergy
* Renal dysfunction (creatinine above normal laboratory limits)
* Symptomatic asthma
* Women who are pregnant or breast-feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share your images with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. The investigators may also share your research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 10 years following article publication.
Access Criteria: Proposals should be directly submitted to woodardp@wustl.edu.

RESULTS

PARTICIPANT FLOW:
Groups:
- PET-cCTA-cFFR: Patients presenting with stable angina and a moderate pretest likelihood for coronary artery disease (CAD) who are already scheduled to undergo invasive coronary catheterization (ICA) for the clinical indication of angina will be recruited to undergo a Coronary CT Angiography (cCTA) examination with Fractional Flow Reserve (FFR) followed immediately by regadenoson stress-rest N-13 Ammonia Positron Emission Tomography (PET) on the same PET/CT scanner. Patients will undergo their clinically scheduled ICA with FFR within 2 weeks of the imaging procedures.
  Patients will receive two single intravenous injections of 10-12 mCi each of the PET radiotracer N-13 Ammonia, one during rest and one during stress. Stress imaging will occur 30-40 minutes prior to rest imaging. Patients will undergo PET/CT imaging immediately post N-13 Ammonia injection.
Period: Overall Study
Arm/Group | PET-cCTA-cFFR
Started | 21
Completed | 20
Not Completed | 1
Not completed — Radiotracer production failed. Patient received an intervention so did not qualify to come back. | 1

BASELINE CHARACTERISTICS:
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Hypertension [Count of Participants; unit: Participants]
  Yes | 19
  No | 2
Smoking [Count of Participants; unit: Participants]
  Yes | 12
  No | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Flow-limiting Coronary Artery Stenosis on CT
Description: CT presence of flow limiting stenosis (≤ 0.8) as determined by CT-FFR in comparison to invasive coronary artery (ICA) FFR. CT-FFR was determined in the following myocardial segments: left anterior descending (LAD), left circumflex (LCx), and right coronary artery (RCA). The number of coronary artery stenoses as determined by CT (CT-FFR ≤ 0.8) was measured.
Time Frame: Day 1 - Day of Scan
Population: One participant did not undergo imaging. Radiotracer production failed. Patient received an intervention so did not qualify to come back.
Measure: Count of Units; unit: Coronary arteries
Units Other Than Participants: Coronary arteries
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
Number analyzed (Coronary arteries) | 60
Coronary arteries | 8

2. Primary Outcome: Association Between Stress Myocardial Blood Flow (MBF) on PET and Coronary Artery Stenosis on CCTA
Description: Association between N-13 Ammonia PET MBF (mL/g/min) during stress and presence or absence of coronary artery stenosis ≥ 50% diameter on CCTA as determined by measurement in each epicardial coronary artery. The MBF values during stress were categorized as normal or abnormal. Normal MBF is defined as >1.8 mL/g/min. MBF and percent diameter stenosis were determined in the following myocardial segments: left anterior descending (LAD), left circumflex (LCx), and right coronary artery (RCA).
Time Frame: Day 1 - Day of Scan
Population: One participant did not undergo imaging. Radiotracer production failed. Patient received an intervention so did not qualify to return for imaging.
Measure: Count of Units; unit: Coronary arteries
Units Other Than Participants: Coronary arteries
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
Number analyzed (Coronary arteries) | 60
Coronary arteries
  Diameter Stenosis ≥50%: number analyzed (Coronary arteries) | 16
  Diameter Stenosis ≥50%: Abnormal MBF Stress | 9
  Diameter Stenosis ≥50%: Normal MBF Stress | 7
  Diameter Stenosis <50%: number analyzed (Coronary arteries) | 44
  Diameter Stenosis <50%: Abnormal MBF Stress | 17
  Diameter Stenosis <50%: Normal MBF Stress | 27
Statistical Analysis 1: Comparison: PET-cCTA-cFFR; Test type: Equivalence — A Fisher's exact test was performed to determine the association between coronary artery stenosis and PET myocardial blood flow (MBF) values during stress. The following myocardial segments were analyzed: left anterior descending (LAD), left circumflex (LCx), and right coronary artery (RCA). Coronary arteries were categorized as coronary arteries with a diameter stenosis ≥50% or <50%. The MBF values during stress were categorized as normal or abnormal. Normal MBF is defined as >1.8 mL/g/min; p = 0.2522, Fisher Exact — The threshold for statistical significance was p = 0.05

3. Secondary Outcome: Correlation of Myocardial Blood Flow (MBF) by PET to Fractional Flow Reserve (FFR) by CT.
Description: Correlation of CT-FFR and N-13 Ammonia PET MBF (mL/g/min) during stress as determined by measurement in each epicardial coronary artery. Values were determined in the following myocardial segments: left anterior descending (LAD), left circumflex (LCx), and right coronary artery (RCA).
Time Frame: Day 1 - Day of Scan
Population: as for outcome 2
Measure: Number; unit: Pearson correlation coefficient (r)
Units Other Than Participants: Coronary arteries
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
Number analyzed (Coronary arteries) | 60
Pearson correlation coefficient (r) | 0.284
Statistical Analysis 1: Comparison: PET-cCTA-cFFR; Test type: Other — A Pearson's Correlation test was performed between PET MFR during stress and CT-FFR by territory; p = 0.028, Pearson's correlation test — The threshold for statistical significance was p = 0.05; A Pearson's Correlation test was performed between PET MFR during stress and CT-FFR by territory

4. Secondary Outcome: CT-Fractional Flow Reserve (CT-FFR) Global
Description: CT-FFR was calculated using a computational flow/AI FFR program (Siemens). Normal CT-FFR was defined as >0.80.
Time Frame: Day 1 - Day of Scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
Ratio
  All Participant Analyzed | 0.90 (0.09)
  Participants with Normal CT-FFR: number analyzed (Participants) | 17
  Participants with Normal CT-FFR | 0.93 (0.05)
  Participants with Abnormal CT-FFR: number analyzed (Participants) | 3
  Participants with Abnormal CT-FFR | 0.73 (0.02)

5. Secondary Outcome: Instant Wave Free Ratio (iFR)
Description: The instant wave Free Ratio (iFR) was measured during the patient's clinically scheduled invasive coronary catheterization. Normal iFR was defined as ≥ 0.90.
Time Frame: Day of invasive coronary catheterization - within 2 weeks of imaging
Population: iFR was done for 8 coronary arteries in 7 participants.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Coronary arteries
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 7
Number analyzed (Coronary arteries) | 8
Ratio | 0.92 (0.05)

6. Secondary Outcome: N-13 Ammonia PET Global Myocardial Blood Flow (MBF) Stress
Description: Myocardial Blood Flow was measured by N-13 Ammonia positron emission tomography (PET) during stress following injection of regadenoson.
Time Frame: Day 1 - Day of Scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
mL/g/min | 1.88 (0.45)

7. Secondary Outcome: N-13 Ammonia PET Global Myocardial Blood Flow (MBF) Rest
Description: Myocardial Blood Flow (MBF) was measured by N-13 Ammonia positron emission tomography (PET) at rest.
Time Frame: Day 1 - Day of Scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
mL/g/min | 0.94 (0.23)

8. Secondary Outcome: N-13 Ammonia PET Global Myocardial Flow Reserve (MFR)
Description: Myocardial flow reserve (MFR) is a ratio between myocardial blood flow (MBF) during stress and at rest, as determined by positron emission tomography (PET). Normal MFR was defined as > 2.0.
Time Frame: Day 1 - Day of Scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PET-cCTA-cFFR
Number analyzed (Participants) | 20
Ratio
  All Participants Analyzed | 2.05 (0.45)
  Participants with Normal MFR: number analyzed (Participants) | 12
  Participants with Normal MFR | 2.31 (0.31)
  Participants with Abnormal MFR: number analyzed (Participants) | 8
  Participants with Abnormal MFR | 1.67 (0.33)

ADVERSE EVENTS:
Time Frame: Within 1-3 days following the imaging procedures and between 25-30 days after invasive coronary artery (ICA) catheterization
Description: Study staff contacted participants by phone following the imaging procedures and invasive coronary artery (ICA) catheterization to confirm the subject's well-being and to ascertain if an adverse event occurred. Subjects received a phone call within 1-3 days following the imaging procedures and between 25-30 days after invasive coronary artery (ICA) catheterization.
Arm/Group | PET-cCTA-cFFR
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
1. Small number of patient subjects.
2. Small number of patients with coronary artery stenoses ≥50% diameter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT05349084/Prot_SAP_000.pdf